CLINICAL TRIAL: NCT01943734
Title: The Influence of Health Information in Stretch Break Program Participant's Lifestyle: a Quantitative and Qualitative Study
Brief Title: The Influence of Health Information in Stretch Break Program Participant's Lifestyle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Caroline de Oliveira Martins, PhD, Federal University of Paraíba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CEPHULW298/09
Record Dates: First submitted 2013-09-10; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Health Behavior
Keywords: Information; Lifestyle; Occupational Health
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle counseling (Experimental): Information passed on anthropometric assessment
  Interventions: Behavioral: Information passed on anthropometric assessment

INTERVENTIONS:
Behavioral: Information passed on anthropometric assessment — Information passed on worker's anthropometric assessment.

SUMMARY:
Objective: To verify the influence of information passed during anthropometric assessment would have in physical exercise (PhE) and eating habits of 14 participants (female=11; 51,07+-8,17 years) from the Stretch Break Program of Federal University of Paraíba (SBP of FUPb). Methods: The research was a descriptive cross-sectional quantitative and qualitative approach. Were applied, between March and May of 2010, anthropometric evaluation and semi-structured interviews. During the evaluation were provided information and guidance on health.

ELIGIBILITY:
Inclusion Criteria:

* FUPb white collar workers of either gender

Exclusion Criteria:

* Anyone who did not complete anthropometric measurements

Ages: 28 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-03; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Anthropometric evaluation | Up to 6 weeks
  Height (cm) was measured with a stadiometer (Sanny), body weight (kg) was measured using a digital scale (TechLine), circumference (cm) was measured (Sanny) at the midpoint between lower costal margin and the superior iliac crest and blood pressure (mmHg) was measured with a sphygmomanometer and a stethoscope (Premium). Direct measurement assessed body mass index, waist-to-height-ratio and blood pressure classification (determined by highest blood pressure category - systolic blood pressure or diastolic blood pressure).

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Martins, PhD, Principal Investigator — Federal University of Paraiba